CLINICAL TRIAL: NCT00432393
Title: Effect of Levodopa-Carbidopa on Visual Function in Patients With Recent-Onset Nonarteritic Anterior Ischemic Optic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8125
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2007-02

CONDITIONS: Nonarteritic Anterior Ischemic Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — carbidopa, levodopa drug combination

INTERVENTIONS:
Drug: levodopa-carbidopa

SUMMARY:
Purpose: There are some controversies about the effect of Levodopa-Carbidopa on treatment of non-arteritic anterior ischemic optic neuropathy (NAION). This study was performed to evaluate the effect of Levodopa-Carbidopa on visual acuity, color vision, and visual field in patients with recent onset NAION (less than 6 weeks duration).

Patients and Methods: In this double-blind randomized clinical trial, 13 patients were treated with levodopa-carbidopa and 12 patients took placebo for 3 weeks. Visual acuity, color vision, and visual field were tested before and at 4th, 12th, 16th, and 24th weeks after enrollment, and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 50 years old
* first ophthalmic examination within 6 weeks after onset of disease
* presence of optic disc swelling followed by optic atrophy within 6 weeks
* altitudinal, central or generalized visual field defect
* normal ESR

Exclusion Criteria:

* confirmed giant cell arteritis
* history of any ocular surgeries
* optic neuropathy due to acute bleeding
* advanced diabetic retinopathy
* uncontrolled glaucoma
* any ocular disorders that cause visual acuity reduction rather than NAION

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Pakravan, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Ophthalmic research center, Tehran, Tehran Province, Iran